CLINICAL TRIAL: NCT06979791
Title: Comparison Between the Effects of Adding Intranasal Dexmedetomidine to Two Different Doses of Midazolam as a Premedication in Pediatrics Undergoing Elective Surgery: A Randomized Controlled Trial
Brief Title: Comparing Two Doses of Midazolam With Added Dexmedetomidine for Kids Before Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed AbdElaty Hamed Ellhwany, Assistant Lecturer, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD-394-2024
Record Dates: First submitted 2025-04-29; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Preoperative Anxiety Experienced by the Pediatric Patient; Preoperative Anxiety
Keywords: "pediatric premedication" "dexmedetomidine" "midazolam" "sedation" "mask acceptance"
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine + Midazolam 0.4 mg/kg (Experimental)
  Interventions: Drug: Dexmedetomidine + Midazolam 0.4 mg/kg
- Dexmedetomidine + Midazolam 0.2 mg/kg (Experimental)
  Interventions: Drug: Dexmedetomidine + Midazolam 0.2 mg/kg

INTERVENTIONS:
Drug: Dexmedetomidine + Midazolam 0.4 mg/kg — Participants in this arm will receive intranasal dexmedetomidine at a dose of 2 mcg/kg combined with intranasal midazolam at a dose of 0.4 mg/kg, administered 30 minutes before the induction of general anesthesia.
  Arms: Dexmedetomidine + Midazolam 0.4 mg/kg
Drug: Dexmedetomidine + Midazolam 0.2 mg/kg — Participants in this arm will receive intranasal dexmedetomidine at a dose of 2 mcg/kg combined with intranasal midazolam at a dose of 0.2 mg/kg, administered 30 minutes before the induction of general anesthesia.
  Arms: Dexmedetomidine + Midazolam 0.2 mg/kg

SUMMARY:
The goal of this this randomized controlled trial is to investigate if adding intranasal dexmedetomidine to two different doses of intranasal midazolam provides effective sedation with fewer side effects in pediatric patients aged 1 to 8 years undergoing elective surgeries. The main questions it aims to answer are:

Does combining intranasal dexmedetomidine with a reduced dose of midazolam achieve adequate sedation while minimizing adverse effects?

How do different dosing regimens affect mask acceptance, parent separation, sedation levels, recovery times, and perioperative adverse events?

Researchers will compare two groups: one receiving dexmedetomidine plus a higher dose of midazolam (0.4 mg/kg) and another receiving dexmedetomidine plus a lower dose of midazolam (0.2 mg/kg) to see if the reduced dose maintains sedation effectiveness while reducing side effects.

Participants will:

Receive intranasal dexmedetomidine (2 mcg/kg) combined with either 0.4 mg/kg or 0.2 mg/kg of intranasal midazolam.

Undergo sedation scoring at 15 and 30 minutes after drug administration.

Be assessed for ease of separation from parents and acceptance of anesthesia mask.

Be monitored for vital signs, recovery times, and any perioperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1 to 8 years
* Scheduled for elective surgery under general anesthesia
* Surgery duration < 1 hour
* ASA physical status I or II
* Parent or legal guardian able to provide informed consent

Exclusion Criteria:

* Refusal to participate by parent/guardian
* Nasal infections, pathology, or epistaxis
* Runny nose or upper respiratory tract infection
* Enlarged adenoids
* BMI > 30
* Known allergy to dexmedetomidine or midazolam
* Fever on day of surgery
* Coagulopathy
* Scheduled for cardiothoracic or neurosurgical procedures
* Congenital heart disease
* Neurological or mental disorders
* Pre-existing sedation (MOASS < 5) on the day of surgery

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mask Acceptance Score (MAS) at time of induction | At the time of induction (approximately 30 minutes after premedication)
  Mask acceptance will be assessed at the time of anesthesia induction using the Mask Acceptance Score (MAS). A score of 1 or 2 will be considered satisfactory (excellent/good), while scores of 3 or 4 will be considered unsatisfactory. The percentage of children with satisfactory mask acceptance will be compared between groups.

SECONDARY OUTCOMES:
Sedation Level (MOASS) at 15 and 30 minutes after premedication | 15 minutes and 30 minutes after drug administration
  Sedation will be evaluated using the Modified Observer's Assessment of Alertness/Sedation Scale (MOASS). Scores will be recorded at 15 and 30 minutes after intranasal drug administration.
Child-Parent Separation Score | Approximately 30 minutes after premedication (at time of separation)
  Measured using the Child-Parent Separation Scale at the time of separation from parents. Scores of 1 or 2 indicate satisfactory separation; score of 3 indicates poor separation.
Heart Rate | Baseline and immediately before anesthesia induction.
  Heart rate will be monitored at baseline and at the time of transfer to the operating room. Mean heart rate values will be compared between the two groups.
Blood Pressure | Baseline and immediately before anesthesia induction
  Mean blood pressure will be monitored at baseline and at the time of transfer to the operating room. Mean blood pressure values will be compared between the two groups.
Time to Recovery (Modified Aldrete Score ≥ 9) | From extubation until Modified Aldrete Score ≥9 is achieved, assessed up to 1 hour in the Post-Anesthesia Care Unit (PACU)
  The time from extubation to achieving a Modified Aldrete Score of ≥9 will be recorded.
Perioperative Adverse Events | From the time of drug administration until 1 hour post-discharge from the Post-Anesthesia Care Unit (PACU), or until the occurrence of a recorded adverse event, whichever comes first.
  Incidence of adverse effects such as nasal irritation, nausea, vomiting, paradoxical reactions, respiratory depression, etc., will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kasr Al-Ainy Hospital, Cairo University, Cairo
  - Souad Kafafi University Hospital, Misr University for Science and, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mountain BW, Smithson L, Cramolini M, Wyatt TH, Newman M. Dexmedetomidine as a pediatric anesthetic premedication to reduce anxiety and to deter emergence delirium. AANA J. 2011 Jun;79(3):219-24. PMID 21751690
- [Background] Cohen LB, Delegge MH, Aisenberg J, Brill JV, Inadomi JM, Kochman ML, Piorkowski JD Jr; AGA Institute. AGA Institute review of endoscopic sedation. Gastroenterology. 2007 Aug;133(2):675-701. doi: 10.1053/j.gastro.2007.06.002. No abstract available. PMID 17681185
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Anttila M, Penttila J, Helminen A, Vuorilehto L, Scheinin H. Bioavailability of dexmedetomidine after extravascular doses in healthy subjects. Br J Clin Pharmacol. 2003 Dec;56(6):691-3. doi: 10.1046/j.1365-2125.2003.01944.x. PMID 14616431
- [Background] Dhiman T, Verma V, Kumar Verma R, Rana S, Singh J, Badhan I. Dexmedetomidine-Ketamine or Dexmedetomidine-Midazolam Nebulised Drug Combination as a Premedicant in Children: A Randomised Clinical Trial. Turk J Anaesthesiol Reanim. 2022 Oct;50(5):380-387. doi: 10.5152/TJAR.2022.21298. PMID 36301288
- [Background] Gomez-Manzano FJ, Laredo-Aguilera JA, Cobo-Cuenca AI, Rabanales-Sotos J, Rodriguez-Canamero S, Martin-Espinosa N, Carmona-Torres JM. Evaluation of Intranasal Midazolam for Pediatric Sedation during the Suturing of Traumatic Lacerations: A Systematic Review. Children (Basel). 2022 Apr 29;9(5):644. doi: 10.3390/children9050644. PMID 35626821